CLINICAL TRIAL: NCT03468933
Title: Intrapleural Tissue Plasminogen Activator and Deoxyribonuclease Therapy Versus Early Medical Thoracoscopy for Treatment of Pleural Infection: A Randomized Clinical Trial
Brief Title: Fibrinolysis Compared to Thoracoscopy for Pleural Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Principal Investigator, Fayez Kheir,MD,MSc, MD, MSc, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1070390
Record Dates: First submitted 2018-03-05; First posted 2018-03-19 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Pleural Infection; Empyema; Pleural Diseases; Parapneumonic Effusion
MeSH Terms: conditions — Empyema; Pleural Diseases | interventions — Tissue Plasminogen Activator; Thoracoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fibrinolytic therapy group (Active Comparator): Patients randomized to the Fibrinolytic group will receive intrapleural therapy of combined tissue plasminogen activator (tPA) and human recombinant deoxyribonuclease (DNase) via chest tube.
  Interventions: Drug: tissue plasminogen activator (tPA) and human recombinant deoxyribonuclease (DNase)
- Medical Thoracoscopy group (Active Comparator): Patients randomized to the Thoracoscopy group will undergo medical thoracoscopy.
  Interventions: Procedure: Medical Thoracoscopy

INTERVENTIONS:
Drug: tissue plasminogen activator (tPA) and human recombinant deoxyribonuclease (DNase) — Patients will receive intrapleural combination of TPA (10 mg) and DNAse (5 mg). Therapy will be given twice daily for a maximum of 6 dose
  Arms: Fibrinolytic therapy group
Procedure: Medical Thoracoscopy — Medical thoracoscopy will be performed as per standard protocols.
  Other Names: Pleuroscopy
  Arms: Medical Thoracoscopy group

SUMMARY:
The purpose of this prospective randomized clinical trial is to compare two currently accepted standard-of-care treatment strategies: Medical thoracoscopy as compared to instillation of intrapleural tissue Plasminogen Activator (TPA) and human recombinant Deoxyribonuclease (DNase) for the management of empyema or complicated parapneumonic effusion (CPPE) in adults.

DETAILED DESCRIPTION:
Background: Pleural infection (empyema or complex parapneumonic effusion (CPPE)) represents one of the most common clinical diagnoses encountered in clinical practice in the United States (US) It is associated with substantial morbidity and mortality despite advances in medical diagnostic and therapeutic strategies.

Objective: Compare two standard of care treatments: TPA/DNase vs early medical Thoracoscopy

Methods: Investigators will conduct a prospective randomized clinical trial. Plan is to enroll total of 32 patients and randomize those patients to either Medical Thoracoscopy group or Fibrinolytic Therapy group.

Follow-up will be daily until hospital discharge and at 6 and 12 weeks in the outpatient setting

Potential Outcome and Benefit: Determine best strategy for treating patients with pleural infection

ELIGIBILITY:
Inclusion Criteria:

Subjects >18 years old with:

Evidence of empyema or complex parapneumonic effusion

Exclusion Criteria:

Age <18 years Pregnancy Inability to give informed written consent Previous thoracic surgery or thrombolytic therapy for pleural infection Medical thoracoscopy cannot be performed within 48 hours Hemodynamic instability or severe hypoxemia Non corrected coagulopathy Homogeneously echogenic effusion on pleural ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fayez Kheir, MD, MSc, Principal Investigator — Tulane University
Locations (1):
- Tulane Medical Center Tulane University Section of Pulmonary DiseasesTulane University Section of Pulmonary Diseases, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fibrinolytic Therapy Group | Medical Thoracoscopy Group
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrinolytic Therapy Group | Medical Thoracoscopy Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [49 to 65] | 65 [62.5 to 72.5] | 64 [54.5 to 69.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 10 | 14 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Ultrasonographic estimated pleural effusion volume,Moderate [Count of Participants; unit: Participants] | 13 | 13 | 26
Number of subjects with community acquired pleural infection [Count of Participants; unit: Participants] | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Duration of Hospital Stay After Intervention
Description: duration of hospital stay in days from time of procedure to discharge from hospital.
Time Frame: 12 week follow up period
Population: All participants received one of the assigned intervention
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fibrinolytic Therapy Group | Medical Thoracoscopy Group
Number analyzed (Participants) | 16 | 16
days | 4 [4 to 5.5] | 2 [2 to 5]

2. Secondary Outcome: Total Length of Hospital Stay
Description: Total days spent in the hospital
Time Frame: 12 week follow up period
Population: All participants received assigned intervention
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fibrinolytic Therapy Group | Medical Thoracoscopy Group
Number analyzed (Participants) | 16 | 16
days | 6 [5 to 8.5] | 3.5 [2 to 10]

3. Secondary Outcome: Number of Participants Necessitating Intervention After the Assigned Treatment
Description: 1. Need for surgical intervention (VATS, Open Thoracotomy) in any arm
  2. Need for additional chest tube and/or fibrinolytic therapy in the medical thoracoscopy arm due to treatment failure
  3. Need of additional chest tube or additional fibrinolytic doses in the fibrinolytic therapy arm due to treatment failure
Time Frame: 12 week follow up period
Population: All participants received assigned intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Fibrinolytic Therapy Group | Medical Thoracoscopy Group
Number analyzed (Participants) | 16 | 16
Participants | 3 | 4

4. Secondary Outcome: Adverse Events
Description: any Adverse events (pain, bleeding)
Time Frame: 12 week follow up period
Population: All participants received assigned intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Fibrinolytic Therapy Group | Medical Thoracoscopy Group
Number analyzed (Participants) | 16 | 16
Participants | 1 | 1

5. Secondary Outcome: In Hospital and 30-day Mortality
Description: Death of a patient while being hospitalized or up to 30 days after
Time Frame: 30 days
Population: All participants received assigned intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Fibrinolytic Therapy Group | Medical Thoracoscopy Group
Number analyzed (Participants) | 16 | 16
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: The perioperative period until hospital discharge, an average of 4 weeks per participant
Description: Definition of adverse event and/or serious adverse event, used to collect adverse event information does not differ from the clinicaltrials.gov.
Arm/Group | Fibrinolytic Therapy Group | Medical Thoracoscopy Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrinolytic Therapy Group (N=16) | Medical Thoracoscopy Group (N=16)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Hemothorax without hemodynamic instability and did not need transfusion, but was monitored in the intensive care unit overnight. Intraprocedural hypoxia that resolved with insertion of a supraglottic airway tube and oxygen therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03468933/Prot_002.pdf
  • Statistical Analysis Plan (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03468933/SAP_003.pdf